CLINICAL TRIAL: NCT00915928
Title: Chronic Subdural Hematoma - Reduction of Recurrence by Treatment With Angiotensin Converting Enzyme Inhibitors
Acronym: KSDH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No effect of the ACE inhibitor evaluated halfway in the study
Sponsor: Odense University Hospital (Other)
Collaborators: Alice Brenaa Foundation (Other); The Hede Nielsen Family Foundation (Other); Overlægerådets legatudvalg (Unknown); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Frantz Rom Poulsen, MD PhD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Chronic Subdural Hematoma; Eudra CT nummer 2009-010058-37
Record Dates: First submitted 2009-06-03; First posted 2009-06-08 (Estimated); Results first posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Hematoma, Subdural, Chronic
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Perindopril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACE inhibitor (Active Comparator): patients randomized to this arm will be treated with ACE inhibitors after surgery
  Interventions: Drug: Perindopril
- Placebo (Placebo Comparator): patients randomized to this arm will be treated with placebo after surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Perindopril — 2,5 mg daily for 3 months
  Other Names: coversyl
  Arms: ACE inhibitor
Drug: Placebo — Placebo dayli for 3 months
  Arms: Placebo

SUMMARY:
The project aims at investigating if treatment with the Angiotensin Converting Enzyme inhibitor Coversyl (perindopril) for 3 months after surgery for chronic subdural hematoma will decrease the risc of recurrence.

DETAILED DESCRIPTION:
Previous studies have indicated that treatment with ACE inhibitors can reduce the risk of recurrence of CSDH after surgical evacuation. This randomized clinical trial was designed to investigate this

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic subdural hematoma that needs surgical evacuation
2. Age > 18 year

Exclusion Criteria:

1. Lack of compliance
2. Kidney artery stenosis
3. Stenosis of the aorta
4. Severely decreased kidney function
5. Allergy or intolerance/contraindications toward ACE inhibitors
6. Already in ACE inhibitor treatment
7. Coagulopathies
8. Malignant disorders
9. Fertile women
10. Other neurological disorders
11. Treatment with pharmaceuticals contraindicating treatment with ACE inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-07; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frantz R Poulsen, MD, PhD, Principal Investigator — Department of Neurosurgery, Odense University Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Neurosurgical clinic
Groups:
- Placebo: Placebo
Period: Overall Study
Arm/Group | ACE Inhibitor | Placebo
Started | 25 | 22
Completed | 25 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with CSDH and indication for surgery. Either male or female
Groups:
- Placebo: three months placebo treatment after surgical CSDH evacuation
- Perindopril: three months perindopril treatment after surgical CSDH evacuation
- Total: Total of all reporting groups
Arm/Group | Placebo | Perindopril | Total
Number analyzed (Participants) | 22 | 25 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (5) | 64.3 (5) | 67.2 (5)
Sex: Female, Male [Count of Participants; unit: Participants] — CSDH and indication for surgical evacuation
  Participants
    Female | 5 | 4 | 9
    Male | 17 | 21 | 38
Region of Enrollment [Number; unit: participants] — Prospective, randomized Population: Many patients were not able to consent and the neurosurgeon on call were too busy to include in the project
  participants
    Denmark | 22 | 25 | 47
Size of Chronic Subdural Hematoma [Mean (Standard Deviation); unit: cm^3] | 130 (10) | 124 (10) | 127 (10)

OUTCOME MEASURES:

1. Primary Outcome: Size of Chronic Subdural Hematoma (CSDH)
Description: Volume of CSDH remnant three months after evacuation measure using xyz/2 on CT scans
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | ACE Inhibitor | Placebo
Number analyzed (Participants) | 25 | 22
cm^3 | 28.4 (5) | 22.8 (5)

2. Secondary Outcome: Composition of Chronic Subdural Hematoma Fluid
Description: Post-Hoc Outcome Measure
Time Frame: years
Population: Analysis will not be performed due to insufficient funding and the samples will be destroyed
Groups:
- Composition of Chronic Subdural Hematoma Fluid: Biochemical analysis of CSDH fluid content. This analysis will not be performed due to insufficient funding
Arm/Group | Composition of Chronic Subdural Hematoma Fluid
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Low dose of a well tolerated and well known drug in the active drug arm
Groups:
- ACE Inhibitor: Active compound
- Placebo: Inactive placebo
Arm/Group | ACE Inhibitor | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/22
Other Adverse Events (participants affected / at risk) | 0/25 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No